CLINICAL TRIAL: NCT05458635
Title: Predictors of Pulmonary Hypertension in Patients With Hypersensitivity Pneumonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Kamal Ibrahim Hassan, Assistant Professor of pulmonology, Cairo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS-131-2019
Record Dates: First submitted 2022-07-04; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension; Hypersensitivity Pneumonitis
MeSH Terms: conditions — Hypertension, Pulmonary; Alveolitis, Extrinsic Allergic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HP without Pulmonary hypertion (No Intervention): HRCT chest , pulmonary functions and echocardiography
- HP with Pulmonary hypertion (Active Comparator): HRCT chest , pulmonary functions ,echocardiography and RT heart catheter in high echocardiographic probability of PH
  Interventions: Procedure: Right heart catheter

INTERVENTIONS:
Procedure: Right heart catheter — Right heart catheterization was performed for 4 cases with high probability of pulmonary hypertension using multi-lumen swan ganz catheter.
  Arms: HP with Pulmonary hypertion

SUMMARY:
Hypersensitivity pneumonitis (HP) is a complex immune mediated disorders caused by repeated inhalation of and sensitization to wide range of antigens including organic particles and chemical compounds, leading to exaggerated immuneresponse. Hypersenstivity pneumonitis is a common form of diffuse parenchymal lung diseases in Egypt .Pulmonary hypertension has been found as a complication of a number of diseases affecting the lung interstitium, including hypersensitivity pneumonitis, with subsequent affection of the life expectancy Rationale of the study: to find predictors for the development of pulmonary hypertension in patients with hypersensitivity pneumonitis

DETAILED DESCRIPTION:
Cross sectional study included 60 patients with established diagnosis of HP , work up includes history of exposure, clinical examination, HRCT chest, ABGs,6MWD, desaturation degree , spirometry, echocardiography and right heart catheter in patients with high echo probability of PH.

ELIGIBILITY:
Inclusion Criteria:

* All patients with confirmed diagnosis of Hypersensitivity pneumonitis

Exclusion Criteria:

* Other interstitial lung diseases

Ages: 29 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of pulmonary hypertension in patients with HP | 6 months
  primary oucome

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy school of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elnady MA, Elkorashy R, Nabil A, Ibrahim EK. Predictors of pulmonary hypertension in patients with hypersensitivity pneumonitis. BMC Pulm Med. 2023 Feb 9;23(1):61. doi: 10.1186/s12890-023-02347-1. PMID 36759788